CLINICAL TRIAL: NCT01797419
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Ranging Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GS-5806 in Subjects < 24 Months of Age Hospitalized for Respiratory Syncytial Virus (RSV) Related Respiratory Infection
Brief Title: Safety Study of GS-5806 to Treat Respiratory Syncytial Virus (RSV)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-218-0104
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory; Syncytial; Virus; RSV
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Virus Diseases | interventions — presatovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GS-5806 (Experimental): Single dose, oral liquid, .5 mL/kg
  Interventions: Drug: GS-5806
- Placebo (Placebo Comparator): Single dose, oral liquid, .5 mL/kg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-5806 — Single dose, oral liquid, .5 mL/kg
  Arms: GS-5806
Drug: Placebo — Single dose, oral liquid, .5 mL/kg
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of GS-5806 in hospitalized infants with RSV.

ELIGIBILITY:
Inclusion Criteria:

* <24 months of age
* Diagnosis of Respiratory Syncytial Virus (RSV) within 48 hours of screening

Exclusion Criteria:

* Chronic or congenital heart disease
* Required ventilation or admission to any pediatric Intensive Care Unit
* Inadequate organ function

Ages: 1 Hour to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 10 days from subject randomization to study drug
  Safety and tolerability will be assessed by evaluating AE's, laboratory abnormalities and vital sign measurements.

SECONDARY OUTCOMES:
Pharmacokinetics effects of GS-5806 | 10 days from subject randomization to study drug
  Evaluation of GS-5806 on viral load related and symptom related endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sly, MD, Principal Investigator — Queensland Children's Medical Research Unit, Herston, AUS
Locations (9):
- Australia (9):
  - Geelong Hospital, Geelong, Victoria
  - Monash Medical Center, Clayton
  - Queensland Children's Medical Research Unit, Herston
  - Royal Hobart Hospital, Hobart
  - Women's and Children's Hospital Adelaide, North Adelaide
  - Royal Children's Hospital, Parkville
  - Sydney Children's Hospital, Randwick
  - Princess Margaret Hospital for Children, Subiaco
  - Westmead Children's Hospital, Westmead